CLINICAL TRIAL: NCT02968082
Title: The Effects of Preoperative Scopolamine Patch Application on the Postoperative Nausea and Vomiting in Microvascular Decompression Surgery
Brief Title: The Effects of Preoperative Scopolamine Patch Application on the Postoperative Nausea and Vomiting in MVD Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung Ho Han, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MVD
Record Dates: First submitted 2016-10-19; First posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Patients
Keywords: MVD; Scopolamine; Microvascular Decompression
MeSH Terms: interventions — Scopolamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo group (P group) (Placebo Comparator): The group that not existed scopolamine ingredient.
  dosage form: apply
  dosage: 1.5 mg
  frequency: 1 times (at 9 p.m. of the day before the operation day)
  duration: Until the 24hr after operation.
  Patients will be applied patch that not existed scopolamine ingredient.
  Interventions: Drug: Placebo
- Scopolamine group (S group) (Experimental): 'Scopolamine (1.5mg) 1 patch'
  The group that existed scopolamine ingredient
  dosage form: apply
  dosage: 1.5 mg
  frequency: 1 times (at 9 p.m. of the day before the operation day)
  duration: Until the 24hr after operation.
  Patients will be applied patch that existed scopolamine ingredient.
  Interventions: Drug: Scopolamine

INTERVENTIONS:
Drug: Scopolamine — Patch will be applied under the ear of the opposite side of operation, at 9 p.m. of the day before the operation day. Nausea will be assessed by Visual Analogue Scale (VAS) immediate after arrival at a recovery room and the ward. After that, nausea will be continuously assessed every 4 hour (4hr, 8hr, 12hr, 16hr, 20hr, and 24hr after surgery) and a number of vomiting will also be counted. Basic clinical characteristics and the number of antiemetic administration will be identified through medical records.
  Arms: Scopolamine group (S group)
Drug: Placebo — Patch will be applied under the ear of the opposite side of operation, at 9 p.m. of the day before the operation day. Nausea will be assessed by Visual Analogue Scale (VAS) immediate after arrival at a recovery room and the ward. After that, nausea will be continuously assessed every 4 hour (4hr, 8hr, 12hr, 16hr, 20hr, and 24hr after surgery) and a number of vomiting will also be counted. Basic clinical characteristics and the number of antiemetic administration will be identified through medical records.
  Arms: Placebo group (P group)

SUMMARY:
A Single-center, randomized, prospective, experimental, double-blind comparison study for effects of preoperative scopolamine patch application on the postoperative nausea and vomiting in microvascular decompression surgery

DETAILED DESCRIPTION:
1. Study design and plan

   1-1) Sixty envelopes will be prepared: Thirty envelopes of scopolamine patch for experimental group and 30 of placebo patch for control group. Each envelope will be tagged for QR code, randomly mixed and numbered from 1 to 60. QR code will be identified after discontinuation of study, so both researchers and subjects would not know in which group the envelope is belonged to.

   1-2) Patch will be applied under the ear of the opposite side of operation, at 9 p.m. of the day before the operation day.

   1-3) Nausea will be assessed by Visual Analogue Scale (VAS) immediate after arrival at a recovery room and the ward. After that, nausea will be continuously assessed every 4 hour (4hr, 8hr, 12hr, 16hr, 20hr, and 24hr after surgery) and a number of vomiting will also be counted. Basic clinical characteristics and the number of antiemetic administration will be identified through medical records.
2. Efficacy assessment

   2-1) Degree of nausea: Visual Analogue Scale (VAS) Subjects will describe their subject degree of nausea by VAS score, just immediate after arrival at a recovery room or the ward and 4hr, 8hr, 12hr, 16hr, 20hr, and 24hr after surgery. Respondents specify their degree of nausea by indicating a point along a continuous 10cm line between two end-points; left one is for "No nausea" and the right one for "Very severe nausea". Scoring is based on the length from left point and higher score means more severe degree of nausea.

   2-2) Number of vomiting Number of vomiting is counted from immediate after arrival at recovery room or the ward, 4hr, 8hr, 12hr, 16hr, 20hr, and 24hr after operation and will be recorded. If there is no vomiting, it will be recorded as "0".

   2-3) Number of antiemetic administration It will be recorded from immediate after arrival at recovery room or the ward, 4hr, 8hr, 12hr, 16hr, 20hr, and 24hr after operation. The kind of antiemetic used and the dosage or number of administration can be identified through medical records.

   2-4) Type of antiemetic and time of administration 2-4-1) PRN) Meckool 10mg/2ml 1amp IVs When VAS is more than 5 or when subjects want at minimum interval of 6hour and maximum of three times. If there is no improvement, it will be noticed.

   2-4-2) PRC) Nasea 0.3mg 1amp IVs
3. Statistical plans

   3-1) General characteristics and clinical characteristics will be analyzed by frequency, percentage, mean value and standard deviation.

   3-2) Homogeneity of variances between experimental group and control group will be analyzed by Chi-square test, t-test and Fisher's exact test 3-3) Degree of nausea between experimental group and control group at recovery room or the ward, 4hr, 8hr, 12hr, 16hr, 20hr, and 24hr after operation will be analyzed by Student's t-test.

   3-4) Number of vomiting and antiemetic administration between experimental group and control group will be analyzed by Fisher's exact test.

   3-5) Hospitalization period between experimental group and control group will be analyzed by Student's t-test.
4. Experimental group of scopolamine patch application will be expected to have less severity of nausea and fewer numbers of vomiting or antiemetic usages. Ultimately, this may relate to hospitalization period and it will be decreased.

ELIGIBILITY:
Inclusion Criteria:

1. Those of either hemi-facial spasm or trigeminal neuralgia, who undergo microvascular decompression (MVD), understand study objectives and voluntarily consent with participation.
2. Adequate communication ability enough to understand and answer the questionnaire.
3. Age ≥ 18 years, and ≤ 65 years.
4. ASA Physical Status Classification from 1 to 2. Class 1: A normal healthy patient Class 2: A patient with mild systemic disease
5. Those who is discharged to general ward, not intensive care unit (ICU) after operation
6. Normal liver or kidney function

Exclusion Criteria:

1. More than one craniotomy in the same period of admission
2. Pregnant or lactating women
3. Narrow-angle glaucoma
4. Pyloric stenosis, intestinal obstruction, bladder obstruction
5. Bradycardia
6. Voiding difficulty such as benign prostate hypertrophy (BPH)
7. Any history of hypersensitivity to ointment base or scopolamine patch

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change in Degree of nausea: Visual Analogue Scale (VAS) | just immediate after arrival at a recovery room or the ward and 4hr, 8hr, 12hr, 16hr, 20hr, and 24hr after surgery
  Subjects will describe their subject degree of nausea by VAS score, just immediate after arrival at a recovery room or the ward and 4hr, 8hr, 12hr, 16hr, 20hr, and 24hr after surgery. Respondents specify their degree of nausea by indicating a point along a continuous 10cm line between two end-points; left one is for "No nausea" and the right one for "Very severe nausea". Scoring is based on the length from left point and higher score means more severe degree of nausea.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Ho Han, PhD, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sato K, Sai S, Adachi T. Is microvascular decompression surgery a high risk for postoperative nausea and vomiting in patients undergoing craniotomy? J Anesth. 2013 Oct;27(5):725-30. doi: 10.1007/s00540-013-1621-9. Epub 2013 May 7. PMID 23649917
- [Background] Pergolizzi JV Jr, Philip BK, Leslie JB, Taylor R Jr, Raffa RB. Perspectives on transdermal scopolamine for the treatment of postoperative nausea and vomiting. J Clin Anesth. 2012 Jun;24(4):334-45. doi: 10.1016/j.jclinane.2011.07.019. PMID 22608591
- [Background] Einarsson JI, Audbergsson BO, Thorsteinsson A. Scopolamine for prevention of postoperative nausea in gynecologic laparoscopy, a randomized trial. J Minim Invasive Gynecol. 2008 Jan-Feb;15(1):26-31. doi: 10.1016/j.jmig.2007.08.616. PMID 18262140
- [Background] Apfel CC, Zhang K, George E, Shi S, Jalota L, Hornuss C, Fero KE, Heidrich F, Pergolizzi JV, Cakmakkaya OS, Kranke P. Transdermal scopolamine for the prevention of postoperative nausea and vomiting: a systematic review and meta-analysis. Clin Ther. 2010 Nov;32(12):1987-2002. doi: 10.1016/j.clinthera.2010.11.014. PMID 21118734